CLINICAL TRIAL: NCT03592030
Title: Diagnostic and Prognostic Value of Miss-1 Study in Children and Adult With Nephrotic Syndrome MISSNEPHROTIQUE
Acronym: MISS-N
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17036
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Nephrotic Syndrome
Keywords: Idiopathic nephrotic syndrome; Minimal change diseases; Primitive FSGS
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The nephrotic syndrome is a rare disease defined by a proteinuria >3g/24h and a hypoalbuminemia < 30g/L. Genetic and immune are the main causes. The acquired idiopathic nephrotic syndrome presents histologically minimal glomerular lesions, sometimes associated with segmental and focal hyalinosis. The idiopathic nephrotic syndrome (INS) represents 85% of children's glomerular nephropathy and 25-30% of adult's.

Relapses are frequents, and can be pejorative up to 10% and lead to end-stage kidney failure.

Another immune cause is the extramembranous glomerulonephritis mediated by molecular targets specific autoantibodies expressed at the podocytes surface.

Other immune causes include lupus nephropathy, ANCA vascularitis, Goodpasture disease, Berger disease.

Easy diagnosis between these causes can be made with the renal biopsy.

Miss-1, a new protein activated during a inflammatory event, could be an actor in nephrotic syndromes by modifying the podocyte's adhesion on the glomerular basal membrane. This would modulate the structure and function of the slit diaphragm, as well as junctions between the podocyte and the glomerular basal membrane, regulating podocytes' apoptosis.

DETAILED DESCRIPTION:
This project is meant to propose and validate specific and non-invasive diagnostic and prognostic tests for the acquired idiopathic nephrotic syndrome.

These tests rely on the measure of Miss-1 expression in circulating blood cells on flow cytometry and its plasmatic concentration.

To date, no equivalent tests exist to diagnose idiopathic nephrotic syndrome (INS) from other causes.

These simple tests would allow a quick diagnosis of acquired INS by avoiding an invasive renal biopsy. It would also help anticipate the relapses of the disease and guide the treatment modalities as do nowadays the PLA2R antibodies in idiopathic membranous nephropathy.

We will propose the tests to every consent patient, hospitalized in the participating centers (Néphrologie pédiatrique of Robert Debré hospital, Néphrologie adulte of Tenon hospital) with a nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All new hospitalized patient
* Presenting a nephrotic syndrome according to its definition
* For which an anatomopathological diagnostic and its evolution can be or will be carried
* Children of any age can be included if they present a nephrotic syndrome

Exclusion Criteria:

- Patients already treated with glucocorticoids and/or immunosuppressor

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All nephrotic patients from the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Miss1 expression in circulating blood cells on flow cytometry at the time of diagnostic of nephrotic syndrome. | From Day 0 to 1 month
  Sensitivity of the Miss1 test: The diagnosis will be made if the expression of Miss1 of circulating leukocytes in flow cytometry at the time of the diagnosis of nephrotic syndrome is> 20 times the mean value of the healthy controls.

SECONDARY OUTCOMES:
Miss1 plasmatic concentration at the time of the diagnostic of nephrotic syndrome | From Day 0 to 1 month
  Sensitivity of plasma Miss1 concentration for INS diagnosis. Specificity, PPV, NPV of the test in the child. Sensitivity, specificity, PPV, NPV of the diagnostic test of the monocyte and granulocyte membrane expression, of lymphocyte subpopulations, Treg and Th17, of the Miss-1 in flow cytometry at the time of the diagnosis of nephrotic syndrome> at a threshold.
Miss1 expression in circulating blood cells on flow cytometry after remission | After remission, up to 1 month
Miss1 plasmatic concentration after remission | After remission, up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Boffa, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Néphrologie et Dialyses Paris, Hôpital Tenon, Paris, France

REFERENCES:
- [Background] Shalhoub RJ. Pathogenesis of lipoid nephrosis: a disorder of T-cell function. Lancet. 1974 Sep 7;2(7880):556-60. doi: 10.1016/s0140-6736(74)91880-7. PMID 4140273
- [Background] Eddy AA, Symons JM. Nephrotic syndrome in childhood. Lancet. 2003 Aug 23;362(9384):629-39. doi: 10.1016/S0140-6736(03)14184-0. PMID 12944064
- [Background] van den Berg JG, Weening JJ. Role of the immune system in the pathogenesis of idiopathic nephrotic syndrome. Clin Sci (Lond). 2004 Aug;107(2):125-36. doi: 10.1042/CS20040095. PMID 15157184